CLINICAL TRIAL: NCT00215761
Title: A Multicenter Study to Investigate Preventive Pacing in Combination With Antiarrhythmic Beta-Blocker Oder AT-I-/ACE-inhibitor Therapy on the Recurrence of Atrial Fibrillation in Patients With Dual-chamber Pacemakers
Brief Title: Recurrence of Atrial Fibrillation in Patients With Dual-chamber Pacemakers and Drug Therapy
Status: Completed | Type: Observational
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: Medtronic BRC (Industry)
Responsible Party: Sponsor
Other Study IDs: AFNET-B05
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Preventive stimulation; Pacemaker
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Comparison of AF-Burden in patients with paroxysmal atrial fibrillation and the necessity of a Dual-Chamber-Pacemaker-Therapy either with a DDD[R]60-Stimulation or AF prevention pacing. All Patients were stratified according to their existing drug therapy, e.g. Beta-Blocker or ACE-Inhibitor.

DETAILED DESCRIPTION:
Implantable pacemaker devices are available with specific atrial pacing algorithms designed to prevent atrial arrhythmias (Preventive stimulation). These algorithms work by increasing the atrial pacing rate to achieve continuous overdrive pacing or by responding to triggers such as premature atrial complexes.

Different investigation's showed that preventive atrial pacing was associated with a 30 to 50 % reduction in the risk of recurrence of AF, compared with no pacing. But a complete recurrence-free long-term effect is not reached.

A hybrid therapy consisting of a combination of preventive atrial stimulation and pharmacologic therapy maybe useful in restoring sinus rhythm. The HOPE-(Heart Outcomes Prevention Evaluation)-Trial showed a overwhelming evidence that, in a broad range of high-risk patients, an ACE-Inhibitor (Ramipril) prevents cardiovascular death, stroke, and heart failure. AF leads to an activation of the renin-angiotensin system (RAS), which seems to play an important role in atrial remodeling. Both experimental and clinical data have confirmed the pro-arrhythmic role of the RAS and demonstrated an anti-arrhythmic effect of ACE- and AT-I-Inhibitors. Madrid et al. showed that a combination of the AT-I-Inhibitor irbesartan plus amiodarone decreased the rate of AF recurrences, with a dose-dependent effect, in AF patients. ACE- and AT-I-Inhibitors represent new and efficient therapeutical options to contrast the nearly inevitable progression of this arrhythmia towards its permanent form. Beta-Blockers are a common pharmacologic therapy in AF patients.

The aim of the BACE-PACE-Trial is to investigate preventive pacing stimulation (PS) vs. standard DDD[R]-60-Stimulation (ST) in combination with antiarrhythmic Beta-Blocker or ACE-inhibitor therapy on the recurrence of atrial fibrillation in patients with dual-chamber pacemakers

The Responder (patients without AF recurrence, respectively with a significant reduction in AF burden) are compared to the standard stimulation. A clinically relevance meant a reduction in AF burden of more than 25 % (experts consensus).

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal symptomatic atrial fibrillation
* Implantation of a dual-chamber pacemaker because of generally accepted pacing indications
* Symptomatic sinus bradycardia, sinus arrest, Tachy-Brady-Syndrome
* Symptomatic sinuatrial block
* Advanced AV-block (AV block II / III)
* Binodal disease: Sick-sinus-syndrome and advanced AV-block
* AV-Nodal-Ablation in combination with pacemaker therapy ( "Ablate & Pace").
* The implantation of a fully functional DDDR Selection 9000, Prevent AF, T 70 DR pacemaker (Vitatron) e.g. normal impedance, stimulation thresholds and sensing values) 2 - 4 months after implantation
* Written informed consent of the patient
* Age > 18 years

Exclusion Criteria:

* Chronic heart failure (NYHA III/IV)
* Acute myocardial infarction < 6 months
* Hypertrophic obstructive cardiomyopathy
* Symptomatic hypo- or hyperthyroidism
* Instable angina pectoris
* Cardiogenic shock
* Patients with diabetes mellitus and recurrent hypoglycaemia
* Pregnancy or breast feeding
* Participation in a clinical trial within the last 30 days. Simultaneous participation in a registry (e.g. project AB1 of the AFNET) is permitted
* Reduced life expectancy (< 6 months)
* Legal incapacity, or other circumstances which would prevent the patient from understanding the aim, nature or extent of the clinical trial
* Evidence of an uncooperative attitude

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paroxysmal symptomatic atrial fibrillation with implemented dual-chamber pacemakers
Sampling Method: Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schuchert, Prof. Dr., Principal Investigator — University Cardiac Center, Hamburg, Germany
Locations (1):
- University Cardiac Center, Hamburg, Hamburg, Germany

REFERENCES:
- See also: German Atrial Fibrillation Network — http://www.kompetenznetz-vorhofflimmern.de